CLINICAL TRIAL: NCT02191020
Title: Multi-center, Randomized, Double Blind, Placebo Parallel-Controlled Study of the Efficacy and Safety of Total Glucosides of Paeony Combined With Acitretin Capsules to Treat Psoriasis Vulgaris
Brief Title: Efficacy and Safety Study of Total Glucosides of Paeony Combined With Acitretin to Treat Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, xjpfW, Chief in Department of Dermatology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XijingH-PF-20120909
Record Dates: First submitted 2014-01-08; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Psoriasis
Keywords: Total Glucosides of Paeony(TGP); Acitretin Capsules; Psoriasis Vulgaris
MeSH Terms: conditions — Psoriasis | interventions — Acitretin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Total glucosides of paeony & Acitretin Capsules (Experimental): During the first week，0.6g，oral，b.i.d.During the other weeks，0.6g，oral，t.i.d
  Interventions: Drug: Total glucosides of paeony & Acitretin Capsules
- Acitretin Capsules (Active Comparator): 20mg/day oral,when subject's weight less than 70kg;otherwise,30mg/day oral.
  Interventions: Drug: Acitretin Capsules

INTERVENTIONS:
Drug: Total glucosides of paeony & Acitretin Capsules
  Arms: Total glucosides of paeony & Acitretin Capsules
Drug: Acitretin Capsules
  Arms: Acitretin Capsules

SUMMARY:
This is a randomized, double blind, placebo parallel-controlled, multi-center clinical trial. Patients with psoriasis vulgaris were randomly divided into the experiment group （treated with TGP combined with acitretin capsules) and control group （treated with placebo combined with acitretin capsules）.The treatment lasted 12 weeks. The efficacy and safety were evaluated at the baseline, as well as 2, 4, 8 and 12 weeks after the beginning of treatment.The investigator's hypothesis TGP combined with Acitretin Capsulesin is more safe and effective than Acitretin Capsulesin to treat Psoriasis Vulgaris.

ELIGIBILITY:
Inclusion Criteria:Meet the following conditions

1. Diagnosed according to Classification criteria for Psoriasis vulgaris;
2. Patients aged 18 to 65 years (to the date of screening);
3. PASI grade>7point<20 point;
4. Not treatment in the Topical corticosteroids、Immunosuppresso、Biologicals agents or Tretinoin cream、Phototherapy nearly one months before enrolled.
5. Understanding the whole process of the study, voluntary participation and signed the informed consent;
6. Patient compliance is good, can guarantee in course of observation.

Exclusion Criteria:One of the following is not included in this study:

1. Pregnant women, ready to pregnant or lactating women;
2. Known to root of herbaceous peony total glycosides (TGP) drug allergy;
3. Have a serious heart, lung, kidney and other vital organs and endocrine system lesions and the history
4. Patients is liver function abnormal persons (ALT above the center laboratory normal limit) or hepatitis b patient grain carriers;
5. Need insulin control of diabetes; High blood pressure did not get good controller ;
6. Patients with white blood cells <4.0 × 109 / L, or a definite anemia (hemoglobin less than 100g / L), or platelets <100 × 109 / L, or other blood disease;
7. Patients with chronic diarrhea, or peptic ulcer nearly 1 year;
8. Patients suffering from malignant tumor;
9. Patients suffering from acute and chronic infectious diseases;
10. Mental disorders, history of alcohol abuse, drug or other substance abuse; 11. Other cases which researchers believe that can not enroll.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Reduction in Psoriasis Area and Severity Index | week 0 and week 12
  After 12 weeks treatment, relative to baseline, the proportion of patients achieving a 50% reduction in Psoriasis Area and Severity Index 50 (PASI50) was 90% in the experiment group and 70.5% in the control group (P<0.05).

SECONDARY OUTCOMES:
incidence of elevated Alanine aminotransferase | week 0 and week12
  After 12 weeks treatment, relative to baseline,the incidence of elevated Alanine aminotransferase (ALT) was 6.8% in the experiment group and 22.2% in the control group (P<0.05).

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospitial, Xi'an, Shaanxi, China